CLINICAL TRIAL: NCT07209579
Title: Evaluation of Mandibular Bone Structure Differences Between Individuals With Periodontitis and Healthy Individuals on Panoramic Radiographs Using Fractal and Morphometric Analyses: A Retrospective Study
Brief Title: Fractal and Morphometric Analysis of Mandibular Bone in Periodontitis
Acronym: PBFM
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Sedef Ayşe Taşyapan, Research Assistant, PhD, Istanbul University
Other Study IDs: 1717821
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Periodontitis; Panoramic Radiography
Keywords: Fractal analysis, Morphometric indices, Panoramic radiography, Mandibular bone, Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Periodontitis Group: Individuals diagnosed with periodontitis based on 2017 EFP/AAP classification
- Healthy Control Group: Systemically and periodontally healthy individuals

SUMMARY:
This retrospective study aims to evaluate the differences in mandibular bone structure between individuals with periodontitis and healthy controls using panoramic radiographs. Fractal analysis and radiomorphometric indices, such as the mental index (MI) and panoramic mandibular index (PMI), will be applied to assess trabecular and cortical bone. The study population includes patients previously diagnosed and treated for periodontitis and healthy individuals with available panoramic radiographs. By comparing bone quality and microarchitecture between the groups, the study seeks to determine the diagnostic value of panoramic radiographs for detecting periodontal bone changes and to provide insights for early diagnosis and treatment planning in dental practice.

DETAILED DESCRIPTION:
Periodontitis is a common inflammatory disease characterized by the destruction of tooth-supporting tissues, often caused by specific microorganisms. In addition to clinical evaluation, radiographic assessment of alveolar bone loss is essential for the diagnosis, treatment planning, and prognosis of periodontal diseases. Panoramic radiography is widely used in oral and maxillofacial imaging and can provide valuable information about cortical and trabecular bone structures through quantitative methods.

Fractal analysis is a mathematical approach that measures the complexity and trabecular patterns of bone. It has been shown to be independent of projection geometry and is commonly applied in digital radiographs. The fractal dimension (FD) reflects the degree of trabecular complexity and can serve as a numerical indicator of bone microarchitecture. The box-counting method, as described by White and Rudolph, will be employed in this study using ImageJ software. In addition to fractal analysis, morphometric indices such as the mental index (MI) and panoramic mandibular index (PMI) will be calculated to assess mandibular cortical thickness and morphology.

This retrospective observational study will include 120 panoramic radiographs obtained from the archives of the Department of Oral and Maxillofacial Radiology, Istanbul University Faculty of Dentistry. The study group will consist of patients with a confirmed diagnosis of periodontitis according to the 2017 classification by the European Federation of Periodontology and the American Academy of Periodontology, while the control group will include systemically healthy individuals with no periodontal disease. Exclusion criteria include individuals under 18 years of age, those with systemic or syndromic conditions, and radiographs with diagnostic errors.

Radiographic measurements will be performed independently by two oral and maxillofacial radiologists, and intra- and inter-observer agreement will be tested through repeated evaluations. Statistical analyses will be conducted using NCSS 2007 software, applying descriptive statistics, Shapiro-Wilk test for normality, independent t-test or Mann-Whitney U test for group comparisons, and chi-square tests for categorical data, with a significance level of p<0.05.

The study is expected to reveal quantitative differences in mandibular bone structure between individuals with periodontitis and healthy controls. The results may contribute to improved diagnostic accuracy of panoramic radiographs in periodontal disease and provide additional tools for early detection and risk assessment in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 or older
* Patients with clinically and radiographically diagnosed periodontitis (case group)
* Periodontally and systemically healthy individuals (control group)

Exclusion Criteria:

* Individuals younger than 18
* Patients with systemic or syndromic conditions affecting bone structure
* Panoramic radiographs with artifacts or diagnostic errors

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consisted of adults aged 18 years and older who underwent panoramic radiographic examinations at the Department of Oral and Maxillofacial Radiology, Istanbul University. The case group included patients diagnosed with periodontitis based on clinical and radiographic criteria, while the control group included periodontally and systemically healthy individuals.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Difference in fractal dimension values between periodontitis and healthy groups | At baseline
  Fractal dimension (FD) values of mandibular bone will be measured from panoramic radiographs using ImageJ software and compared between periodontitis patients and healthy controls.

SECONDARY OUTCOMES:
Differences in morphometric indices between groups | At baseline
  Morphometric indices will be calculated and compared between periodontitis patients and healthy controls.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Faculty of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No